CLINICAL TRIAL: NCT00003249
Title: A Phase I Investigation of Carboxyamido-triazole (CAI) Modulated by Ketoconozole In Patients With Advanced Malignancies
Brief Title: Carboxyamidotriazole and Ketoconazole in Treating Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02265; UCCRC-9019; NCI-T97-0086; CDR0000066129 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — carboxyamido-triazole; Drug Therapy; Ketoconazole

ARMS (1):
- Arm I (Experimental): Patients receive oral carboxyamidotriazole (CAI) as a test dose on day 1. Patients receive oral ketoconazole on day 7, followed by CAI plus ketoconazole on day 8. CAI and ketoconazole are administered in combination on day 1 and days 3-28 of the first course. Ketoconazole is administered alone on day 2 of the first course. Subsequent courses begin at 28 day intervals in the absence of disease progression or unacceptable toxic effects. Cohorts of 3 patients are evaluated at each dose level prior to dose escalation. If one of three patients within a cohort experiences dose limiting toxicity (DLT), that dose level is expanded to incorporate six patients. If two or more patients experience DLT, the next lower dose is declared to be the maximum tolerated dose.
  Interventions: Drug: carboxyamidotriazole; Drug: chemotherapy; Drug: ketoconazole

INTERVENTIONS:
Drug: carboxyamidotriazole
Drug: chemotherapy
Drug: ketoconazole

SUMMARY:
Phase I trial to study the effectiveness of carboxyamidotriazole and ketoconazole in treating patients with advanced cancers. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of carboxyamidotriazole (CAI) in combination with ketoconazole in patients with advanced malignancies.

II. Evaluate the toxic effects, safety, and efficacy of CAI in combination with ketoconazole.

III. Determine the modulatory effects of ketoconazole on the pharmacokinetic profile of CAI.

IV. Determine a pharmacodynamic model for CAI and ketoconazole with respect to potential gastrointestinal, hematologic, and neurotoxicities.

OUTLINE: This is a dose escalation study.

Patients receive oral carboxyamidotriazole (CAI) as a test dose on day 1. Patients receive oral ketoconazole on day 7, followed by CAI plus ketoconazole on day 8. CAI and ketoconazole are administered in combination on day 1 and days 3-28 of the first course. Ketoconazole is administered alone on day 2 of the first course. Subsequent courses begin at 28 day intervals in the absence of disease progression or unacceptable toxic effects. Cohorts of 3 patients are evaluated at each dose level prior to dose escalation. If one of three patients within a cohort experiences dose limiting toxicity (DLT), that dose level is expanded to incorporate six patients. If two or more patients experience DLT, the next lower dose is declared to be the maximum tolerated dose.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven refractory or recurrent nonhematologic malignancies
* Measurable or evaluable disease by radiographic or clinical examination

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance Status: Karnofsky 70-100%
* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT no greater than 2.5 times upper limit of normal
* Albumin at least 3 g/dL
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance greater than 60 mL/min
* No concurrent neurotoxicities greater than grade 1 from previous chemotherapy
* No concurrent neuropathy greater than grade 1
* Not pregnant
* Effective contraceptive method must be used by fertile patients during and up to 2 months after study
* No serious uncontrolled medical illness
* No history of active inflammatory bowel disease, ileus, or other chronic malabsorption syndromes

PRIOR CONCURRENT THERAPY:

* No concurrent isoniazid
* No concurrent rifampin
* At least 4 weeks since chemotherapy
* At least 6 weeks since nitrosoureas therapy
* At least 3 months since suramin therapy
* No prior carboxyamidotriazole
* No concurrent steroids (except dose required for adrenal insufficiency)
* No concurrent tamoxifen
* No prior radiotherapy within 4 weeks of study
* No prior total gastrectomy or total ileocolectomy
* No concurrent therapy with H2 antagonists, barbiturates, calcium channel blockers, terfenadine, astemizole, cisapride, digitoxin, quinidine, amiodarone, carbamazepine, imipramine, or antacids
* No concurrent erythromycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-05; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Ratain, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States